CLINICAL TRIAL: NCT02580539
Title: A Phase I/II Open-label Study of the Safety and Efficacy of Epstein-Barr Virus Specific T-cell Lines for the Treatment of EBV Infection or EBV-related Lymphoproliferative Diseases
Brief Title: A Study of the Safety and Efficacy of EBV Specific T-cell Lines
Acronym: EBV-TCL-01
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dr. Jean-Sebastien Delisle, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Dr. Jean-Sebastien Delisle, MD, PhD, Clinician-Scientist, Hematopoietic Cell Transplantation Program, Maisonneuve-Rosemont Hospital
Organization: Maisonneuve-Rosemont Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CER15020
Record Dates: First submitted 2015-10-15; First posted 2015-10-20 (Estimated); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Epstein-Barr Virus Infections; Post-Transplant Lymphoproliferative Disorder; Lymphoma
Keywords: Allogeneic Transplantation; T cell; Epstein-Barr Virus
MeSH Terms: conditions — Epstein-Barr Virus Infections; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Autologous or allogenic (stem cell donor) T cells (Experimental): Subjects receive an autologous anti-EBV T-cell line or a T-cell line derived from the patient's allogeneic (stem cell transplant) donor.
  Interventions: Biological: Group A
- Allogeneic "third party" T cells (Experimental): Subjects receive a T-cell line from a matched or partially matched related donor.
  Interventions: Biological: Group B

INTERVENTIONS:
Biological: Group A — Peptide-stimulated T cells 2 x 10^7/m^2
  Arms: Autologous or allogenic (stem cell donor) T cells
Biological: Group B — Peptide-stimulated T cells per dose-escalation protocol
  Arms: Allogeneic "third party" T cells

SUMMARY:
This study evaluates the safety and efficacy of EBV-specific T-cell lines to treat patients suffering from high EBV viral titers not responding to standard of care therapies and to treat EBV-related lymphoma. The study will recruit 6 patients to receive autologous T cells or a T cell line derived from the patient's allogeneic donor (in the case of stem cell transplant recipients), and 6 patients to receive a T-cell line prepared from a matched or partially matched related donor.

DETAILED DESCRIPTION:
Epstein-Barr virus (EBV) is a member of the herpes virus family and infects up to 95% of individuals over their lifetime. Most initial infections occur in childhood and after a brief flu-like illness, the virus enters a phase of latency.

Patients who receive a bone marrow transplant or an organ transplant take medications drugs that weaken their immune systems. In these contexts, the virus can "reactivate" and cause very serious problems, such as lymphoma. For unknown reasons, people with a normal immune system can also develop lymphoma due to EBV.

The purpose of this study is to test the safety and efficacy of immune cells (T lymphocytes) that are specifically "taught" to recognize the virus-infected cells and to eliminate them. This "education" occurs is done over during a 2 weeks period (approximately), in the research laboratory. The cells are then transfused into the patient.

ELIGIBILITY:
Inclusion Criteria:

* Capacity to provide informed consent
* Age ≥ 18 years old
* Confirmed treatment-refractory EBV reactivation or EBV-related lymphoma
* ECOG of 2 or less

Exclusion Criteria:

* Medical condition requiring a corticosteroid dose greater than Prednisone 0.5mg/kg/day (or equivalent) at the time of the infusion.
* Patient has received T-cell depleting antibodies or stem cell transplantation in the 28 days prior to proposed date of anti-EBV T-cell line infusion
* Patient has received a solid organ transplant in the 3 months prior to proposed date of anti-EBV T-cell line infusion.
* Pregnant or nursing females
* Life expectancy of less than 3 months due to a condition unrelated to the EBV- related disease.
* Active uncontrolled GVHD
* Active uncontrolled SOT rejection episode

DONOR ELIGIBILITY: An allogeneic donor must be a first-degree relative with at least 3/6 HLA compatibility, have consented to donate peripheral blood mononuclear cells, and fulfill the same criteria for stem cell donation according to the hospital's standard operating procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2015-11; Primary Completion 2025-05 (Actual); Study Completion 2025-05 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence and description of CTCAE v.4.03 adverse events related to the experimental treatment | During observation period (up to 42 days post infusion)
  Complications: infusional toxicity, immune-related and other

SECONDARY OUTCOMES:
Changes in EBV titers (viral load) for each patient | Until 12 months post infusion
  As measured by PCR weekly until week 6, at 3 months, 6 months and 12 months
Immune reconstitution as measured by various laboratory assays of immune cell type and function | During observation period until 12 months post infusion
  ELISpot on peripheral blood is assessed at the time points mentioned above
All cause mortality | At 12 months
  Within the 12 months observation period
Transplant-related outcomes | During observation period until 12 months post infusion
  Incidence/severity of graft-versus-host disease, solid organ rejection episodes, relapse
Incidence/severity of graft-versus-host disease among patients who underwent stem cell transplantation | During observation period until 12 months post infusion
  Based on standardized assessments done weekly until week 6 and at 3, 6 and 12 months
Number and severity of solid organ rejection episodes per patient among those who underwent solid organ transplant | During observation period until 12 months post infusion
  Based on standardized assessments done weekly until week 6 and at 3, 6 and 12 months
Incidence of primary disease relapse among patients who underwent stem cell transplantation | During observation period until 12 months post infusion
  Based on standardized assessments done weekly until week 6 and at 3, 6 and 12 months
Malignancy staging for patients with lymphoma, per internationally-accepted guidelines for the different specific lymphomas | During observation period until 12 months post infusion
  As clinically indicated by the investigators and/or primary physician

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Sebastien Delisle, MD,PhD, Principal Investigator — Maisonneuve-Rosemont Hospital
Locations (1):
- Hôpital Maisonneuve-Rosemont, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Center for Excellence in Cell Therapy — https://ciusss-estmtl.gouv.qc.ca/propos/axes-dexcellence/therapie-cellulaire